CLINICAL TRIAL: NCT05868642
Title: Impatto Emodinamico Dell'Anestesia Subaracnoidea Titrata Nel Confronto Con la Tecnica Tradizionale Single-shot Nei Pazienti Sottoposti ad Artroprotesi d'Anca. Trial Randomizzato Controllato
Brief Title: Impatto Emodinamico Dell'Anestesia Subaracnoidea Titrata Versus Tecnica Single-shot Nei Pazienti Sottoposti ad Artroprotesi d'Anca. RCT
Acronym: NINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0000440
Record Dates: First submitted 2018-05-13; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia; Adverse Effect; Anesthesia, Local
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T group (Experimental): Subaracnhoid block levobupivacaine 0.5%, 10 mg (2 ml) via subarachnoid injection plus 1mg for each metameric level needed to achieve the T10 level sensory block (evaluation with pinprick test at 10 minute after the firts injection and at 4 minute from the second injection)
  Interventions: Procedure: subarachnoid block
- S group (Active Comparator): levobupivacaine 0.5%, 15 mg (3 ml) via subarachnoid injection
  Interventions: Procedure: subarachnoid block

INTERVENTIONS:
Procedure: subarachnoid block — subarachnoid block with levobupivacaine at different dosage for pation undergoing total hip arthroplasty

SUMMARY:
Studying the hemodynamic effects of titrated subarachnoid anesthesia versus conventional single-shot subarachnoid anesthesia

DETAILED DESCRIPTION:
This study aims to investigate whether a different hemodynamic effect is related to the injection o titrated local anesthetic for subarachnoid anesthesia versus the conventional single shot injection. The data to be recorded are blood pressure and pulse rate at different timing. As secondary outcomes the investigators will record the anesthetic level achieved using the Bromage score.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-40 kg/m2
* ASA 1-3
* undergoing total hip arthroplasty
* no controindications to subaracnhoid block
* able to understand and sign a written informed consensus
* METs > o = 4

Exclusion Criteria:

* baseline SBP < 100 mmHg

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
SBP change | 60 minute
  SBP will be recorded at baseline and every 5 minutes after the subarachnoid block for 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: battista borghi, professor, Principal Investigator — isituto ortopedico rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy